CLINICAL TRIAL: NCT01539850
Title: Safety Evaluation of the LGL102 in Obese Subjects Treated With OMS102. A Prospective Multicenter Study
Brief Title: Safety Evaluation of the LGL102 in Obese Subjects Treated With OMS102
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IntraPace, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-006
Record Dates: First submitted 2012-02-22; First posted 2012-02-28 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Obesity; Morbid Obesity
Keywords: obesity; gastric stimulation; morbid obesity
MeSH Terms: conditions — Obesity; Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: OMS102 — Subjects will receive implanted OMS102 System.
  Other Names: abiliti System

SUMMARY:
The main objective of this study is to evaluate the LGL102 implant safety in obese to morbidly obese subjects treated with OMS102 system. The effect of the therapy on body weight changes will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 - 60 years old at time of screening
* BMI of 35 to 55 at time of screening
* History of obesity ≥ 5 years
* The subject has been under routine care of the investigator or another single physician that can supply a medical record for at least 6 months prior to enrollment
* Women with childbearing potential (i.e., not post-menopausal or surgically sterilized) must agree to use adequate birth control methods
* No significant weight loss (< 5%) within four months prior to enrollment as documented in the subject's medical record.
* Successful psychological evaluation following the institution psychological evaluation protocol for bariatric surgery or successful historic assessment performed no more than 6 months prior to enrollment.
* Glycosylated Hemoglobin; HbA1c ≤ 7.0 % at Visit 2 or historic value performed no more than 3 months prior to enrollment.
* If taking anti-depressant medications, they must be stable for at least six months prior to enrollment
* Willingness to refrain from using prescription, over the counter or herbal weight loss products for the duration of the trial
* Alert, mentally competent, and able to understand and willing to comply with the requirements of the clinical trial, and personally motivated to abide by the requirements and restrictions of the clinical trial
* Able to provide voluntary informed consent

Exclusion Criteria:

* Any prior bariatric surgery
* Other implanted electrical stimulation devices (e.g. pacemaker, defibrillator, neurostimulator)
* Diagnosed with past or current psychiatric condition that may impair his/her ability to comply with the study procedures
* Use of anti-psychotic medications
* Diagnosed with a eating disorder such as bulimia or binge eating
* Obesity due to an endocrinopathy (e.g. Cushing disease)
* Insulin therapy
* GI disease such as hiatal hernia (> 5cm), gastroparesis, esophageal motility disorders or intractable constipation.
* Any history of peptic ulcer disease within 5 years prior to enrollment
* History of Barrett's esophagus
* Women who are pregnant, lactating or anticipate becoming pregnant within 24 months
* Arthritis or other pathologies limiting physical activities that physician feels should exclude the patient from the study.
* Cardiac history that physician feels should exclude the patient from the study.
* Use of another investigational device or agent in the 30 days prior to enrollment
* A history of life-threatening disease within 5 years prior to enrollment
* Any other condition that, in the opinion of the investigator, would make the subject unsuitable for the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2010-03; Primary Completion 2011-04 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Transgastric sensor site healing | 3 months
  Food sensor transgastric site healing will be evaluated during a gastro endoscopy exam performed three months after implant.

SECONDARY OUTCOMES:
Excess weight loss | 3, 6, and 12 months
  Percentage of excess body weight loss (%EWL) compared to baseline.
Safety Evaluation | 3, 6, and 12 months
  Occurrence and severity of all adverse events
Quality of Life | 3, 6 and 12 months
  Evaluation of the quality of life using the Moorehead-Ardelt II questionnaire
Eating Behavior | 3, 6 and 12 months
  Eating behavior (cognitive restraint, uncontrolled eating, and emotional eating) using the Three Factor Eating Questionnaire (TFEQ)
Comorbid Conditions | 3, 6 and 12 months
  Any reduction of blood pressure and oral diabetes medications

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Horbach, MD, Principal Investigator — Stadtkrankenhaus Schwabach
Locations (3):
- Germany (3):
  - Wolfart Klinik, Gräfelfing
  - Stadtkrankenhaus Schwabach, Schwabach
  - Chirurgische Klinik und Poliklinik I Zentrum für Operative Medizin, Würzburg

REFERENCES:
- [Derived] Horbach T, Thalheimer A, Seyfried F, Eschenbacher F, Schuhmann P, Meyer G. abiliti Closed-Loop Gastric Electrical Stimulation System for Treatment of Obesity: Clinical Results with a 27-Month Follow-Up. Obes Surg. 2015 Oct;25(10):1779-87. doi: 10.1007/s11695-015-1620-z. PMID 25771794